CLINICAL TRIAL: NCT06464159
Title: New Therapeutic Strategy Against Preeclampsia : Angiogenic Switch to Physiological State by Extracorporeal Removal of sFlt-1 and Release of PlGF
Brief Title: New Therapeutic Strategy Against Preeclampsia
Acronym: APHERESE2
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP231772; 2023-A01545-40 (Other: ID-RCB)
Record Dates: First submitted 2024-06-03; First posted 2024-06-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Preeclampsia
Keywords: Preeclampsia; Apheresis; Angiogenic factors; Maternal biomarkers; sFLt-1; PIGF; Placenta; Pregnancy
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, serum, plasma, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Preeclampsia: Pregnancy with preeclampsia
  Interventions: Biological: Biological collection
- Pregnancies with intra uterine growth restriction (IUGR): Pregnancy with intra uterine growth restriction (IUGR)
  Interventions: Biological: Biological collection
- Normal pregnancy: Pregnancy without preeclampsia and intra uterine growth restriction (IUGR) and complications
  Interventions: Biological: Biological collection

INTERVENTIONS:
Biological: Biological collection — A collection of maternal plasma, serum and urine

SUMMARY:
Preeclampsia is a hypertensive disorder of pregnancy associated with important maternal and perinatal mortality. It complicates 2 to 5% of pregnancies and causes more than 70 000 maternal deaths each year worldwide. Although symptomatic management has improved there is currently no curative treatment, and only childbirth and delivery of the placenta, usually prematurely, alleviate the mother's symptoms. The management of extremely preterm infants is a major societal challenge in medical, ethical and economic terms.

Placental insufficiency plays a central role in the pathophysiology of preeclampsia. Abnormal placentation during the first trimester leads to placental hypoperfusion, which induces trophoblast dysfunction and the release in maternal circulation of trophoblastic factors leading to the maternal symptoms. Among molecules that participate to the pathophysiology of preeclampsia, one of the most important players is soluble fms-like tyrosine kinase 1 (sFlt-1), which is a soluble form of the vascular endothelial growth factor (VEGF) and placenta growth factor (PlGF) receptor. sFlt-1 binds to free VEGF and PlGF in the maternal circulation, thus reducing their bioavailability for their membrane receptors. Targeting the sFlt-1 pathway is one of the most promising strategies for the development of new treatments for preeclampsia. As sFlt-1 results from alternative splicing, its peptide sequence is identical to that of the extracellular part of the membrane receptor. The development of drugs that act specifically on the soluble form and not on the membrane form is therefore particularly complex.

The general objective of this research is to restore the angiogenic balance that maintains the physiological concentrations of free angiogenic factors in order to significantly prolong the pregnancy and diminish the consequences of the great prematurity. The precise objectives of the APHERESE 2 project are:

1. To transpose the proof of concept of the APHERESE1 project to the scale of a real apheresis column
2. To develop an innovative assay technology to determine the global circulating angiogenic balance for each patient

DETAILED DESCRIPTION:
The aim of this biobank is to setup a collection of maternal plasma and serum from patients with preeclampsia and patients with normal pregnancy. Assays of circulating angiogenic and anti-angiogenic factors (free and total forms) will be carried out on these serum and plasma at the hormonology laboratory in Cochin hospital (Paris, France) These results will make it possible to optimize and validate the development of extracorporeal sFlt-1 purification techniques.

Preeclampsia is a very heterogeneous disease in its clinical presentation, our hypothesis is that this heterogeneity corresponds to different profiles of angiogenic balance disturbance. Not all patients are likely to have the same expected benefit from extracorporeal clearance of sFlt-1. The objective is to assess the overall angiogenic balance on a large number of patients in order to determine which profile best corresponds to the indication for apheresis.

A prospective non-interventional study will be initiated to collect maternal blood samples during normal pregnancies and during pregnancies complicated by preeclampsia (Port-Royal Maternity, Cochin APHP). Blood samples will be collected after collection of written informed consent from 50 patients with preeclampsia and 50 patients without hypertensive disease.

* Between 20WG and 23WG+6D : 10 patients with PE and 10 patients with NP
* Between 24WG and 27WG+6D : 10 patients with PE and 10 patients with NP
* Between 28WG and 31WG+6D : 10 patients with PE and 10 patients with NP
* Between 32WG and 35WG+6D : 10 patients with PE and 10 patients with NP
* Between 36WG and 40WG+6D : 10 patients with PE and 10 patients with NP Inclusion of the patients will be performed through the Cochin maternal/neonatal investigation center.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 50 years old
* Singleton pregnancies between 20 and 41 weeks of gestation
* Preeclampsia / normal pregnancy

Exclusion Criteria:

* Age < 18 years old
* Infectious disease: HIV, HBV or HCV
* Multiple pregnancies
* refusal to participate in the protocol
* Lack of social security cover

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: pregnancy with preeclampsia or intra uterine growth restriction (IUGR) and without preeclampsia and intra uterine growth restriction (IUGR) and complications
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Concentration of total sFlt-1 | 6 months
  in pg/mL - to assess main angiogenic factors during PE, intra uterine growth restriction (IUGR) and normal pregnancy
Concentration of free PlGF | 6 months
  in pg/mL - to assess main angiogenic factors during PE, intra uterine growth restriction (IUGR) and normal pregnancy

SECONDARY OUTCOMES:
Concentration of total PIGF | 6 months
  in pg/mL - to assess global circulating angiogenic balance during PE, intra uterine growth restriction (IUGR) and normal pregnancy
Concentration of total VEGFA | 6 months
  in pg/mL - to assess global circulating angiogenic balance during PE, intra uterine growth restriction (IUGR) and normal pregnancy
Concentration of total sVEGFR2 | 6 months
  in pg/mL - to assess global circulating angiogenic balance, total VEGFA and total sVEGFR2 during PE, intra uterine growth restriction (IUGR) and normal pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Vassilis TSASARIS, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Edouard LECARPENTIER, MD, PhD, Study Chair — Institut National de la Santé Et de la Recherche Médicale, France; Jean GUIBOURDENCHE, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Maternité Port-Royal, Paris, France

IPD SHARING:
Plan to Share IPD: No